CLINICAL TRIAL: NCT06463015
Title: Evaluation of the Effectiveness of Ultrasound-guided Posterior Tibial Nerve Pulsed Radiofrequency Therapy in the Management of Diabetic Neuropathic Pain
Brief Title: Posterior Tibial Nerve PRF for Diabetic Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTNPRF for Diabetic Neuropathy
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Neuropathies, Painful; Diabetic Neuropathy Peripheral
Keywords: Pulsed Radiofrequency Treatment; Ultrasonography; Tibial Nerve
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulsed radiofrequency group (Other): posterior tibial nerve pulsed radiofrequency for painful DPNP
  Interventions: Procedure: ultrasound-guided posterior tibial nerve pulsed radiofrequency

INTERVENTIONS:
Procedure: ultrasound-guided posterior tibial nerve pulsed radiofrequency — The posterior tibial nerve (PTN) was identified with a 5-12 MHz linear ultrasonography (US) probe at the level of the medial malleolus, where it runs posterior to the posterior tibial artery. Using the in-plane technique, a 22-gauge, 10-cm radiofrequency cannula was inserted under US guidance and advanced until the tip was adjacent to the nerve. Pulse radiofrequency was applied at 42°C for 240 s with a pulse width of 20 ms

SUMMARY:
This study aimed to evaluate the efficacy of ultrasound (US)-guided posterior tibial nerve pulsed radiofrequency (PTN PRF) in the treatment of painful diabetic peripheral neuropathy (DPNP) refractory to conservative treatments. For this evaluation, the visual analog scale (VAS), PainDETECT neuropathic pain scores, and Jenkins Sleep Scale (JSS) will be used before and after the PTN PRF.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPNP) is a common complication of diabetes and is observed in approximately 50% of people with diabetes throughout their lives. Approximately 50% of patients complain of neuropathic pain. Diabetic neuropathic pain significantly reduces the quality of life, increases 10-year mortality, and is the main reason why patients seek medical attention. Diabetes affects the peripheral nervous system in various ways, with distal symmetric polyneuropathy being the most common. Patients with distal symmetric polyneuropathy typically complain of progressive unpleasant sensory sensations that are most prominent at night. These sensations may present as tingling (paresthesia), burning pain, electric shock, stabbing pain, pain triggered by contact with clothing and bedding (allodynia), or frostbite-like pain radiating upward from the feet. More than 70% of patients with DPNP have persistent moderate to severe pain, resulting in insomnia, impaired quality of life, and mood disorders. Diabetic neuropathic pain incurs five times more healthcare costs than diabetes itself. International guidelines recommend duloxetine, amitriptyline, pregabalin or gabapentin as first-line agents for symptomatic analgesic treatment in patients with DPNP. However, the response to medical treatment may not always be adequate, or treatment with these drugs may cause many side effects, such as balance disorder, sedation, and weight gain, especially in older patients with comorbidities. The susceptibility of patients with DPNP to drug side effects, comorbidities, and drug-drug interactions results in maximum doses of first-line drugs that are not tolerated. Combination therapies (e.g., Duloxetine + Pregabalin) are known to be more effective in terms of both pain efficacy and patient tolerability compared to high-dose monotherapy. However, comorbidities, drug-drug interactions, and side effects in patients with diabetic peripheral neuropathy who cannot tolerate even the optimum doses of combination therapy are a very serious problem that the physician managing the treatment should overcome. In addition to pharmacological treatments, interventional treatment modalities are also available for patients with DPNP. These methods include spinal cord stimulation (SCS), lumbar sympathetic chain radiofrequency ablation/neurolysis, and dorsal root ganglion stimulation. Invasive methods, such as SCS, are costly and may cause serious complications, such as visceral organ damage and bleeding. Therefore, new treatment options are needed. For this reason, we planned to apply pulse radiofrequency (PRF) treatment to the bilateral posterior tibial nerve (PTN) in patients with TYPE-2 diabetes with painful DPNP to provide a minimally invasive treatment method with limited drug-drug interaction and long-term well-being.

PRF delivers short bursts of high-voltage electrical current to the target nerve, creating a nonthermal effect that modulates the transmission of pain signals. The mechanism of action of PRF is not fully understood, but it is believed to involve changes in synaptic transmission, gene expression, and modulation of inflammatory mediators without causing significant thermal damage or coagulation necrosis to nerve fibers. The PTN is a branch of the sciatic nerve that provides sensory and motor innervation to the heel and the sole of the foot. The advantage of the PTN over its smaller branches is that it can be visualized and targeted using US. While there are a limited number of studies in the literature on interventional procedures in the management of DPNP, no study has evaluated the effectiveness of PRF applied to PTN.

The primary aim of this study was to evaluate the efficacy of PTN PRF treatment for DPNP using VAS and PainDETECT scoring. The secondary aims were to determine the incidence of adverse events associated with US-guided PTN PRF and to evaluate the effect of PTN PRF treatment on sleep quality. A total of at least 51 patients will be enrolled. VAS, painDETECT and Jenkins Sleep Scale (JSS) scores will be assessed pre-treatment, 1 month and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* >5 years of Type 2 DM diagnosis,
* >2 years of neuropathic pain complaints (pain-DETECT score >19),
* Between the ages of 18-70,
* >1 year of persistent severe pain with a VAS>6 despite effective multiple medical treatment,
* Diagnosis of distal symmetric polyneuropathy confirmed by electroneuromyelography (ENMG)

Exclusion Criteria:

* Other diseases that may lead to distal symmetric polyneuropathy (non-DM endocrinopathies, such as B12-folate deficiency),
* Pregnancy
* Coagulopathy, antiaggregant/anticoagulant/antiplatelet use,
* Psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Change from baseline to 1st and 3rd month after treatment
  Visual analog scale (VAS) is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
painDETECT neuropathic pain questionnaire | Change from baseline to 1st and 3rd month after treatment
  The painDETECT questionnaire, is a screening tool designed to identify neuropathic pain components in patients with chronic pain. The unabbreviated name is "painDETECT questionnaire". The score ranges from 0 to 38, with higher scores indicating a greater likelihood of neuropathic pain. Higher scores mean a higher likelihood of neuropathic pain and a worse poor outcome. A total score of 19 or more is indicative of likely neuropathic pain.
The Jenkins Sleep Scale | Change from baseline to 1st and 3rd month after treatment
  The Jenkins Sleep Scale (JSS) is a scale used to measure sleep quality. The JSS consists of four items related to common sleep problems: difficulty falling asleep, waking up several times during the night, difficulty staying asleep, and waking up tired. It uses a Likert-type scale ranging from 0 to 5, where 0 represents "not at all" and 5 corresponds to "22-31 days." The total JSS score is the sum of four items, with a range from 0 (no sleep problems) to 20 (most sleep problems). Higher scores indicate more acute sleep difficulties. Therefore, in this context, higher scores on the JSS reflect worse sleep outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Yildiz, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)